CLINICAL TRIAL: NCT00004343
Title: Study of Hypercortisolism in Cushing's Syndrome and Stress-Induced Pseudo-Cushing's Syndrome
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: Oregon Health and Science University (Other)
Other Study IDs: NCRR-M01RR00334-0028; OHSU-3324
Record Dates: First submitted 1999-10-18; First posted 1999-10-19 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2003-12

CONDITIONS: Cushing's Syndrome
Keywords: Cushing's syndrome; endocrine disorders; rare disease
MeSH Terms: conditions — Cushing Syndrome; Endocrine System Diseases; Rare Diseases

SUMMARY:
OBJECTIVES:

I. Determine whether Cushing's syndrome and stress-induced pseudo-Cushing's syndrome can be differentiated by evaluating endogenous corticotropin-releasing hormone activity.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: Patients undergo a 30-hour infusion of deuterated cortisol with peripheral and petrosal vein measurements of adrenocorticotropin hormone (ACTH) and corticotropin-releasing hormone (CRH). Patients also have a 2-day, low-dose dexamethasone suppression test.

Patients with ACTH tumors are referred for pituitary surgery as indicated. Patients without Cushing's syndrome are entered as controls. During scheduled radiologic procedures, these subjects undergo ACTH and CRH sampling from the petrosal vein or cavernous sinus following a deuterated cortisol infusion.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

Suspected adrenocorticotropin hormone (ACTH)-dependent Cushing's syndrome No pregnant women Effective contraception required of fertile women

Min Age: 0 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40
Dates: Start 1999-10

CONTACTS AND LOCATIONS:
Overall Officials: Mary H. Samuels, Study Chair — Oregon Health and Science University
Locations (1):
- Oregon Health Sciences University, Portland, Oregon, United States